CLINICAL TRIAL: NCT03600155
Title: A Phase I Study of Nivolumab in Combination With Ipilimumab for the Treatment of Patients With High Risk or Refractory/Relapsed Acute Myeloid Leukemia and Myelodysplastic Syndrome Following Allogeneic Stem Cell Transplantation
Brief Title: Nivolumab and Ipilimumab After Donor Stem Cell Transplant in Treating Patients With High Risk Refractory or Relapsed Acute Myeloid Leukemia or Myelodysplastic Syndrome
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2017-0349; NCI-2018-01450 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2017-0349 (Other: M D Anderson Cancer Center); P30CA016672 (NIH)
Record Dates: First submitted 2018-07-16; First posted 2018-07-26 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Allogeneic Hematopoietic Stem Cell Transplantation Recipient; Myelodysplastic Syndrome; Recurrent Acute Myeloid Leukemia; Refractory Acute Myeloid Leukemia
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia, Myeloid, Acute | interventions — Ipilimumab; CTLA-4 Antigen; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A (nivolumab) (Experimental): Beginning at least 6 weeks post-stem cell transplant, patients receive nivolumab IV over 60 minutes on days 1 and 15. Treatment repeats every 28 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Nivolumab
- Arm B (ipilimumab) (Experimental): Beginning at least 6 weeks post-stem cell transplant, patients receive ipilimumab IV over 90 minutes on day 1. Treatment repeats every 21 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Ipilimumab
- Arm C (nivolumab and ipilimumab) (Experimental): Beginning at least 6 weeks post-stem cell transplant, patients receive nivolumab IV over 60 minutes on days 1, 14, and 28, and ipilimumab IV over 90 minutes on day 1. Treatment repeats every 6 weeks for up to 6 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Ipilimumab; Biological: Nivolumab

INTERVENTIONS:
Biological: Ipilimumab — Given IV
  Other Names: Anti-Cytotoxic T-Lymphocyte-Associated Antigen-4 Monoclonal Antibody; BMS-734016; MDX-010; MDX-CTLA4; Yervoy
  Arms: Arm B (ipilimumab); Arm C (nivolumab and ipilimumab)
Biological: Nivolumab — Given IV
  Other Names: BMS-936558; MDX-1106; NIVO; ONO-4538; Opdivo
  Arms: Arm A (nivolumab); Arm C (nivolumab and ipilimumab)

SUMMARY:
This phase Ib trial studies the side effects and best dose of nivolumab and ipilimumab after donor stem cell transplant in treating patients with high risk acute myeloid leukemia or myelodysplastic syndrome that does not respond to treatment or has come back. Immunotherapy with monoclonal antibodies, such as nivolumab and ipilimumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose (MTD) and dose limiting toxicity (DLT) of nivolumab and ipilimumab alone and in combination in patients with high risk or refractory/relapsed acute myeloid leukemia (AML) and myelodysplastic syndrome (MDS) following allogeneic stem cell transplantation (allo-SCT).

II. To evaluate the toxicity of nivolumab and ipilimumab alone and in combination with regard to the rate and severity of acute graft versus host disease (aGVHD).

SECONDARY OBJECTIVES:

I. To determine the overall response rate (ORR) of nivolumab, ipilimumab and the combination in patients with high risk or refractory/ relapsed AML and MDS following allo-SCT.

II. To determine the duration of response, disease-free survival (DFS), and overall survival (OS) of patients with high risk or refractory/ relapsed AML and MDS treated with this combination following allo-SCT.

EXPLORATORY OBJECTIVES:

I. To identify neo-antigens, the immune cell phenotype, expression of immune checkpoint molecules and the T cell receptor (TCR) repertoire following treatment with nivolumab, ipilimumab and the combination.

II. To study immunological and molecular changes in the peripheral blood and bone marrow in response to nivolumab and ipilimumab.

III. To investigate the TCR repertoire and immune phenotype in patients who experience aGVHD.

OUTLINE: This is a dose-escalation study. Patients are assigned to 1 of 3 arms.

ARM A: Beginning at least 6 weeks post-stem cell transplant, patients receive nivolumab intravenously (IV) over 60 minutes on days 1 and 15. Treatment repeats every 28 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity.

ARM B: Beginning at least 6 weeks post-stem cell transplant, patients receive ipilimumab IV over 90 minutes on day 1. Treatment repeats every 21 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity.

ARM C: Beginning at least 6 weeks post-stem cell transplant, patients receive nivolumab IV over 60 minutes on days 1, 14, and 28, and ipilimumab IV over 90 minutes on day 1. Treatment repeats every 6 weeks for up to 6 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up within 30 days and periodically thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients with evidence of relapsed or refractory AML or MDS following allogeneic stem cell transplantation
* Patients must have received preparative regimens to include either busulfan- or melphalan-based regimens
* Patient must have achieved myeloid engraftment as defined by an absolute neutrophil count >= 500 micro/L on 3 consecutive days
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Total bilirubin =< 2 times upper limit of normal (x ULN) (=< 3 x ULN if considered to be due to Gilbert's syndrome)
* Aspartate aminotransferase or alanine aminotransferase =< 2.5 x ULN
* Serum creatinine =< 2 x ULN or glomerular filtration rate (GFR) >= 50
* Patients must provide written informed consent
* The interval from the infusion of stem cells to time of initiation of nivolumab or ipilimumab will be at least 6 weeks (42 days)
* Females must be surgically or biologically sterile or postmenopausal (amenorrheic for at least 12 months) or if of childbearing potential, must have a negative serum or urine pregnancy test within 72 hours before the start of the treatment
* Women of childbearing potential must agree to use an adequate method of contraception during the study and until 3 months after the last treatment. Males must be surgically or biologically sterile or agree to use an adequate method of contraception during the study until 3 months after the last treatment

Exclusion Criteria:

* Patients with known allergy or hypersensitivity to nivolumab or ipilimumab or any of their components
* Patients with acute GVHD > grade 2 at any time during the post-transplant course
* Patients with a known history of severe interstitial lung disease or severe pneumonitis or active pneumonitis that is uncontrolled in the opinion of the treating physician
* Patients with a known history of any of the following autoimmune diseases are excluded:

  * Patients with a history of inflammatory bowel disease (including Crohn's disease and ulcerative colitis)
  * Patients with a history of rheumatoid arthritis, systemic progressive sclerosis (scleroderma), systemic lupus erythematosus, autoimmune vasculitis (e.g., Wegener's granulomatosis)
* Patients with solid organ allografts (such as renal transplant) are excluded
* Ongoing immunosuppressive therapy for the treatment of GVHD. Patients receiving GVHD prophylaxis will be allowed on this study
* Patients with symptomatic central nervous system (CNS) leukemia at the time of evaluation or patients with poorly controlled CNS leukemia
* Active and uncontrolled disease/(active uncontrolled infection, uncontrolled hypertension despite adequate medical therapy, active and uncontrolled congestive heart failure New York Heart Association [NYHA] class III/IV, clinically significant and uncontrolled arrhythmia) as judged by the treating physician
* Patients with known human immunodeficiency virus seropositivity will be excluded
* Known to be positive for hepatitis B by surface antigen expression. Known to have active hepatitis C infection (positive by polymerase chain reaction or on antiviral therapy for hepatitis C within the last 6 months)
* Any other medical, psychological, or social condition that may interfere with study participation or compliance, or compromise patient safety in the opinion of the investigator
* Patients unwilling or unable to comply with the protocol
* Pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2018-10-11 (Actual); Primary Completion 2024-12-02 (Actual); Study Completion 2024-12-02 (Actual)

PRIMARY OUTCOMES:
Optimal dose of nivolumab in combination with ipilimumab | Up to day 42
  Dose-finding will be carried out using the Bayesian optimal interval design.

SECONDARY OUTCOMES:
Overall response rate (ORR) | Up to 1 year
  ORR will be estimated as the proportion of patients who achieve complete response (CR), complete response with incomplete bone marrow recovery (CRi), or partial response (PR). The 2-sided 95% exact binomial confidence interval (CI) of ORR will be calculated.
Duration of response (DOR) | From the date of initial response (PR or better) to the date of first documented disease progression/relapse or death, assessed up to 1 year
  DOR will be estimated using the method of Kaplan and Meier, and distributions will be compared using the log-rank test.
Disease-free survival (DFS) | From the date of first dose of study drug until the date of documented graft versus host disease (GVHD), relapses from CR, or death from any cause, assessed up to 1 year
  DFS will be estimated using the method of Kaplan and Meier, and distributions will be compared using the log-rank test.
Overall survival (OS) | From the first dose of study drug until death or last follow-up, assessed up to 1 year
  OS will be estimated using the method of Kaplan and Meier, and distributions will be compared using the log-rank test.

OTHER OUTCOMES:
Neo-antigen identification | Up to 1 year
  Will be detected using McNemar tests or generalized linear mixed model (GLMM).
Immune cell phenotype | Up to 1 year
  Will be detected using McNemar tests or GLMM.
Immune checkpoint molecule expression | Up to 1 year
  Will be detected using McNemar tests or GLMM.
T cell repertoire (TCR) | Up to 1 year
  Will be detected using McNemar tests or GLMM.
Immunological and molecular changes in peripheral blood and bone marrow | Baseline up to 1 year
  Paired t-tests or GLMM will be used.
TCR repertoire in patients who experience acute (a)GVHD | Up to 1 year
  Will be detected using McNemar tests or GLMM.
Immune phenotype in patients who experience aGVHD | Up to 1 year
  Will be detected using McNemar tests or GLMM.

CONTACTS AND LOCATIONS:
Overall Officials: Gheath Al-Atrash, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2023-02-13): https://cdn.clinicaltrials.gov/large-docs/55/NCT03600155/ICF_001.pdf